CLINICAL TRIAL: NCT06504030
Title: A Single-arm, Single-center, Prospective Study of Modified DEP Regimens (Doxorubicin+ Etoposide + Methylprednisolone) for the Treatment of Hemophagocytic Lymphohistiocytosis
Brief Title: Modified DEP Regimens for the Treatment of Hemophagocytic Lymphohistiocytosis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Xuefeng He, Dr, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: modified-DEP
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Hemophagocytic Lymphohistiocytoses
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- modified-DEP for HLH (Experimental): modified-DEP for the treatment of non-EBV-HLH and EBV-HLH patients.
  Interventions: Drug: modified-DEP

INTERVENTIONS:
Drug: modified-DEP — For non-EBV-HLH patients: Liposomes doxorubicin, 25 mg/m2 d1, etoposide 100 mg/m2 d1, methylprednisolone 1 mg/kg d1-3, then tapering according to patients condition, fully stop with d7 to d10; ruxolitinib, 15 mg bid. Emapalumab, if needed.
  For EBV-HLH patients: PD-1 monoclonal antibody, 2 mg/kg (maximum dose, 200 mg) d-3, liposomes doxorubicin, 25 mg/m2 d1, etoposide 100 mg/m2 d1, methylprednisolone 1 mg/kg d1-3, then tapering according to patients condition, fully stop with d7 to d10; ruxolitinib, 15 mg bid. Emapalumab, if needed.

SUMMARY:
This study is trying to evaluate the efficacy and safety of modified DEP regimens for the treatment of active hemophagocytic lymphohistiocytosis.

DETAILED DESCRIPTION:
In the investigators' previous clinical practice, it has been found that under the condition of combined treatment with safer inflammatory factors such as ruxolitinib and CCRT, further reducing the dosage of high-dose hormones and shortening the duration of use can effectively reduce the occurrence of adverse reactions while still achieving the effect of effectively alleviating HLH. This study is a prospective clinical study aimed at observing the effectiveness and safety of the modified DEP regimen in the treatment of active HLH.

ELIGIBILITY:
Inclusion Criteria:

1. According to the HLH-2004 criteria, the patient meets the HLH diagnosis.
2. 1 year old < age < 70 years old, regardless of gender.
3. Before the start of the study, total bilirubin ≤ 10 times the upper limit of normal; serum creatinine ≤ 1.5 times the normal value; fibrinogen can be corrected to ≥ 0.6g/L after infusion.

3. Serum HIV antibody negative; HCV antibody negative, or HCV antibody positive, but HCV-RNA negative. HBV surface antigen and HBV core antibody are both negative. If any of the above is positive, peripheral blood hepatitis B virus DNA titer detection is required, and it must be less than 1×103 copies/ml before enrollment.

4. Women of childbearing age must be confirmed to be non-pregnant through pregnancy tests, and are willing to take effective contraceptive measures during the trial and within ≥ 6 months after the last dose; pregnant and lactating women cannot participate; all male subjects take contraceptive measures during the trial and within ≥ 3 months after the last dose.

5. Sign the informed consent form.

Exclusion Criteria:

1. Allergic to liposome doxorubicin, etoposide, and ruxolitinib or with severe allergic constitution;
2. Severe myocardial damage, with myocardial enzyme CK and CK-MB increased more than 3 times ULN (upper limit of normal value).
3. Patients with heart disease of grade II or above (including grade II) according to the New York Heart Association (NYHA) score.
4. Subjects who have used a total cumulative dose of doxorubicin ≥300mg/m2 or a total cumulative dose of epirubicin ≥450mg/m2, or who have previously used anthracyclines to cause heart disease.
5. Subjects with severe mental illness;
6. Severe and uncontrollable infections, such as lung infection, intestinal infection, and sepsis.
7. Active massive bleeding in visceral organs (including gastrointestinal bleeding, alveolar bleeding, intracranial bleeding, etc.);
8. Patients who are unable to rely during the trial and/or follow-up stage and who are participating in other clinical studies at the same time.

   * For patients who intend to use PD-1 monoclonal antibodies, if the patient has any of the following conditions, PD-1 monoclonal antibodies will not be used, and only the DEP regimen that does not contain PD-1 monoclonal antibodies will be used:

     1. Those who are allergic to PD-1 monoclonal antibody components.
     2. Abnormal thyroid function.
     3. Those who have other severe immune reaction tendencies, including immune myocardial injury, immune hepatitis, immune pneumonia, etc.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Response rate of modified-DEP | 2 weeks, 4 weeks, 6 weeks, 8 weeks
  Rates of complete response, partial response, improvement
Incidence of Treatment-Emergent Adverse Events | 2 weeks, 4 weeks, 6 weeks, 8 weeks
  Rates of adverse events

SECONDARY OUTCOMES:
Survival of patients | 3 months, 6 months, 1 year
  The disease outcomes, 3-month and 6-month survival rates, and median survival

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng He, Dr, Principal Investigator — The First Affiliated Hospital of Soochow University

IPD SHARING:
Plan to Share IPD: Undecided